CLINICAL TRIAL: NCT04946734
Title: Effectivity and Safety of PFO Closure vs Medicine in Alleviating Migraine （SPRING）: a Multicenter, Random, Case Control Study
Brief Title: Effectivity and Safety of PFO Closure vs Medicine in Alleviating Migraine
Acronym: SPRING
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Caojin, MD, Principal Investigator, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPRING2021
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: PFO - Patent Foramen Ovale; Migraine
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders | interventions — Aspirin; Clopidogrel; Tryptamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Arm (Experimental): Device PFO closure
  Interventions: Device: PFO closure device; Drug: Aspirin and clopidogrel; Drug: Triptans
- Control Arm (Other): Drugs only
  Interventions: Drug: Aspirin and clopidogrel; Drug: Triptans

INTERVENTIONS:
Device: PFO closure device — Device PFO closure.
  Arms: Test Arm
Drug: Aspirin and clopidogrel — Aspirin 100mg qd for 6 months and clopidogrel 75mg qd administered for 1month after device implanted.
Drug: Triptans — If migraine recurred, Triptans would be administered during the acute phase.

SUMMARY:
Effectivity and safety of PFO closure vs medicine in alleviating migraine （SPRING）: a multicenter, random, case control study

ELIGIBILITY:
Inclusion Criteria:

1. Presence of PFO with right-to-left shunt, confirmed by Transthoracic.
2. Echocardiography (TTE) or transesophageal echocardiography (TEE) with a bubble study.
3. Bubble study positive confirmed by transcranial doppler.
4. Subject is diagnosed of migraine.
5. Subject signs an informed Consent Form and is willing to participate in follow-up visits

Exclusion Criteria:

1. Subject is diagnosed of headache with clear etiology.
2. Subject had cerebral hemorrhage, bleeding events in other organs within 3 months or was in high risk of bleeding.
3. Brain CT/MR showed ischemic lesions.
4. Subject is diagnosed of hepatic insufficiency: ALT or AST>3×ULN at the screening visit.
5. Subject is diagnosed of moderate to severe renal insufficiency: eGFR<30ml/min/1.73m2 at the screening visit.
6. Subject has uncontrolled arrhythmia with clinical significance within 90 days.
7. Subject is diagnosed of unstable angina, severe coronary atherosclerosis or myocardial infarction within 90 days.
8. Subject is diagnosed of pulmonary artery embolism, peripheral artery embolism or deep Vein Thrombosis.
9. Subject cannot follow the study procedure due to other acute or chronic diseases.
10. Subject is pregnant or lactating.
11. Subject is under other RCT.
12. Subject has a life expectancy <1 year.
13. Subject cannot follow the study procedure due to other reasons in the opinion of the investigators.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
Complete cessation of migraine | Month 12
  Primary Efficacy Endpoint
Serious Adverse Event (SAE) related due to device, drug or study procedure | Month 12
  Primary Safety Endpoint

SECONDARY OUTCOMES:
Monthly migraine attacks | Baseline and Month 12
  Mean change of monthly migraine attacks
Monthly migraine days | Baseline and Month 12
  Mean change of monthly migraine days. Monthly migraine days = migraine attacks in one month × average time period per attacks (hours) /24 hours
Responder rate | Baseline and Month 12
  Percentage of subject with at least 50% reduction in monthly migraine attacks from baseline

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Sanjiu Brain Hospital, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou First People's Hospital, Huizhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - Shangqiu First People's Hospital, Shangqiu, Henan
  - Enshi Huiyi Hospital of Rheumatic Diseases, Enshi, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Zhongnan hospital of wuhan university, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - China-Japan Friendship Hospital of Jilin University, Changchun, Jilin
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The Eighth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Shenzhen
  - The people's hospital of Leshan, Leshan, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
The deidentified participant data will be shared on a request basis.

REFERENCES:
- [Derived] Zi-Yang Y, Hezhi L, Dongling L, Ximeng W, Caojin Z; SPRING Investigators. Rationale and design of the SPRING trail: effectivity and safety of Pfo closuRe vs medIcine in alleviatiNg migraine, a multicenter, randomized and open-label trail. BMC Cardiovasc Disord. 2024 Apr 5;24(1):198. doi: 10.1186/s12872-024-03866-3. PMID 38580946